CLINICAL TRIAL: NCT00816959
Title: Phase III Randomized, Multi-center Study to Evaluate the Effect of R-mabHDI in Patients With Lymphocytic Predominant Hodgkin's Lymphoma
Brief Title: Study Evaluating the Effect of R-mabHDI in Lymphocytic Predominant Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: American Scitech International (Other)
Collaborators: Eli Lilly and Company (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Ratna Grewal MD., American Scitech International
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASI-HDIII 0109
Record Dates: First submitted 2009-01-05; First posted 2009-01-06 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Hodgkin's Lymphoma
Keywords: Lymphocytic Predominant Hodgkin's Lymphoma; Late, widespread and recurrent LPHD
MeSH Terms: conditions — Hodgkin Disease | interventions — ABVD protocol; Doxorubicin; Bleomycin; Vinblastine; Dacarbazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I: R-mabHDI and ABVD (Active Comparator)
  Interventions: Drug: R-mabHDI and ABVD
- Arm II: ABVD (Active Comparator)
  Interventions: Drug: ABVD

INTERVENTIONS:
Drug: R-mabHDI and ABVD — The subjects will receive R-mabHDI intravenously, separately for about 7 hours on days 1,8,15 and 22 (once a week) of every cycle. Each cycle is 4 weeks. R-mabHDI will be given for 2 cycles.
  Also the subjects will receive the ABVD combination intravenously for about 1 hour on day 1 and 15 of every cycle (every 2 weeks). Each cycle is 4 weeks. ABVD will be given for 6 cycles.
  Other Names: R-mabHDI
  Arms: Arm I: R-mabHDI and ABVD
Drug: ABVD — The subjects will receive the ABVD combination intravenously for about 1 hour on day 1 and 15 of every cycle (every 2 weeks). Each cycle is 4 weeks. ABVD will be given for 6 cycles.
  Other Names: Adriamycin, Bleomycin, Vinblastine and Dacarbazine
  Arms: Arm II: ABVD

SUMMARY:
Objective:

The primary objective of the study is to evaluate the effect of R-mabHDI in patients with late stage, widespread stage and recurrent Lymphocytic Predominant Hodgkin's Lymphoma.

The hypothesis is that the combination of R-mabHDI with the standard ABVD therapy in patients with late stage (Stage III and Stage IV) and recurrent stage Lymphocytic Predominant Hodgkin's Lymphoma will have a favorable outcome on the response and progress free survival. The study is also aimed at evaluating the safety of R-mabHDI .

The aim of the study is to test this hypothesis by evaluating the clinical outcome in 1200 patients receiving combination of R-mabHDI once a week for 8 weeks and ABVD therapy every other week for 12 treatments.

DETAILED DESCRIPTION:
The primary objective of the study is to evaluate the effect of R-mabHDI in Patients with late stage, widespread stage and recurrent Lymphocytic Predominant Hodgkin's Lymphoma.

The hypothesis is that the combination of R-mabHDI with the standard ABVD therapy in patients with late stage (Stage III and Stage IV) and recurrent stage Lymphocytic Predominant Hodgkin's Lymphoma will have a favorable outcome on the response and progress free survival. The study is also aimed at evaluating the safety of R-mabHDI .

A total of 1200 subjects will be recruited to the study from various centers. Enrollment period will last for up to one and half year and treatment period is for six months. Treatment will be considered a failure if the tumor size and signs of LPHD does not decrease after 3 months.

Subjects having late stage HD, widespread HD or recurrent HD fulfilling the inclusion and exclusion criteria will be recruited in this study. Females who are nursing babies or are pregnant will be excluded from the study.

All subjects will receive the drugs according to the randomization process. The eligible subjects will be randomly assigned to 1 of 2 "treatment" groups after screening. No matter which group the subjects are assigned to, the doses of the drugs will be the standard doses that are currently used to treat lymphoma.

Group 1: subjects assigned to group 1 will receive the ABVD combination intravenously for about 1 hour on day 1 and 15 of every cycle (every 2 weeks). Each cycle is 4 weeks. ABVD will to be given for 6 cycles.

The subjects will also receive R-mabHDI intravenously, separately for about 7 hours on days 1,8,15 and 22 (once a week) of every cycle. Each cycle is 4 weeks. R-mabHDI will be given for 2 cycles.

Group 2: subjects assigned to group 2 will receive the ABVD combination intravenously for about 1 hour on day 1 and 15 of every cycle (every 2 weeks). Each cycle is 4 weeks. ABVD will to be given for 6 cycles.

Subjects in group 2 will not receive R-mabHDI .

ELIGIBILITY:
Inclusion Criteria:

* Must sign the informed consent form
* Patients with proven diagnosis of Lymphocytic Predominant Hodgkin's Lymphoma in late stage HD, widespread HD and recurrent HD on histology.
* Patients of both gender
* Patients between ages of 16 and 65 years
* Patients must have bi-dimensionally measurable disease
* Patients with adequate bone marrow reserve (ANC>1500/mm3 ; Platelets> 50,000/ mm3)
* LVEF >/= 50% as measured by echocardiogram
* Serum creatinine < 2mg/dl
* Serum bilirubin < 2mg/dl; AST or ALT < 2x ULN
* International Prognostic Score of >2 (Patients must have > 2 of the following risk features: Male >/= 45 years of age, Stage IV, Albumin <4, WBC >/= 15, Lymphocytes < 8% or < 600, Hb < 10.5)

Exclusion Criteria:

* Classic Hodgkin's disease
* Known HIV infection
* Pregnant women and women of child bearing capacity, tests positive on a urine/blood pregnancy test, is lactating/nursing, has had three or more days of amenorrhea at the time of first dose of the treatment, is contemplating pregnancy in next six months or is not using an efficient contraceptive method.
* Severe pulmonary disease as judged by the Principal Investigator including COPD and asthma
* Acute infection requiring treatment with intravenous therapy
* Presence of CNS lymphoma
* Concomitant malignancies or previous malignancies within the last 5 years
* Active Hepatitis B or C infection
* Uncontrolled active infection
* Concurrent prednisone or systemic steroid therapy

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1200 (Estimated)
Dates: Start 2011-07; Primary Completion 2014-04 (Estimated); Study Completion 2014-04 (Estimated)

PRIMARY OUTCOMES:
The primary efficacy criterion is the response rates (RR) by Kaplan-Meier at 3,6,12, and 18 months. | 18 months

SECONDARY OUTCOMES:
Additional secondary endpoint criterion is the progress free survival (PFS) by Kaplan-Meier at 18 months. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Ratna Grewal, MD., Study Chair — American Scitech International- eCRO; Sarath Babu, MD., Principal Investigator — MedCenter Primary and Internal Medicine
Locations (1):
- MedCenter, East Brunswick, New Jersey, United States